CLINICAL TRIAL: NCT01290328
Title: Epoetin Alfa in the Treatment of Post-Transplant Anemia: A Randomized Controlled Trial
Brief Title: Study of Epoetin Alfa to Treat Anemia After Kidney Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment, termination of funding
Sponsor: Mehrotra, Anita, M.D. (Individual)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Anita Mehrotra MD, Principal Investigator, Mehrotra, Anita, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0843; EPONAP2001 (Other Grant/Funding Number: Centocor Ortho Biotech)
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2012-07

CONDITIONS: Anemia
Keywords: anemia; kidney transplant; alloimmunity
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (No Intervention)
- Epoetin alfa (Experimental): 150 units/kg/week
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa — 150 units/kg/weekly
  Other Names: Procrit
  Arms: Epoetin alfa

SUMMARY:
The primary purpose of this study is to determine the effect of Epoetin Alfa (Procrit) on the change in hemoglobin (red blood cell count) in anemic kidney transplant recipients. The investigators hypothesize that epoetin alfa will raise hemoglobin.

DETAILED DESCRIPTION:
Anemia has become an increasingly recognized problem in kidney transplant recipients, and erythropoietin is often prescribed as treatment despite limited data regarding outcomes. Multiple clinical trials have demonstrated correction of anemia with erythropoietin in patients with chronic kidney disease (pre-transplant) and patients on dialysis. No large clinical trials of erythropoietin treatment have been done in anemic kidney transplant recipients, however. The investigators hypothesize that when used for the treatment of post-transplant anemia, Epoetin Alfa increases hemoglobin (Hb). The investigators further hypothesize that Epoetin Alfa suppresses pathogenic alloimmunity directed at the kidney transplant and as a consequence, prevents immune-mediated injury and thereby preserves renal function. Finally, the investigators hypothesize that treatment of post-transplant anemia with Epoetin Alfa also results in improved patient-reported outcomes (quality of life) and decreased left ventricular mass. In order to test these hypotheses, the investigators propose a randomized controlled trial of Epoetin Alfa in anemic kidney transplant recipients (9.0 < Hb < 11.0). 100 study subjects will be randomized to either treatment with Epoetin Alfa at a starting dose of 150 units/kg/week or no treatment (50 subjects/arm). The primary outcome of change in Hb will be measured by CBC at 6 weeks, 3 months, 6 months, and 1 year of enrollment. Secondary outcomes to be measured include change in renal function (eGFR), change in T cell phenotype, change in patient-reported outcomes (SF-36 form), and change in left ventricular mass (by cardiac MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Kidney transplant recipient at least 8 weeks post-transplant
3. Mild to moderate anemia, defined as 9.0 g/dL < Hb < 11 g/dL)
4. Estimated GFR (by MDRD) < 60 mL/min (not on dialysis)
5. Transferrin saturation > 20% and Ferritin > 100 ng/mL

Exclusion Criteria:

1. History of erythrocyte-stimulating agent (ESA) use in the previous 8 weeks
2. Red blood cell transfusion in previous 30 days
3. History of HIV/AIDS
4. Nonfunctioning graft, defined as patient requiring chronic dialysis
5. Hypersensitivity to ESAs or albumin
6. Uncontrolled hypertension, defined as screening BP > 180/100
7. New-onset seizures (diagnosed within the last 3 months) or seizure disorder uncontrolled on medications (breakthrough seizures on medication)
8. History of any neoplasm except: adequately treated basal or squamous cell carcinoma of the skin, solid tumors (except primary CNS lymphoma) treated with curative therapy and disease-free for more than 5 years.
9. Pregnancy or lactating
10. Vitamin B12 deficiency (Vit B12 < 180 pg/mL)
11. Untreated folate deficiency (folate < 6.6 ng/mL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
change in hemoglobin | 6 weeks to 1 year
  The primary outcome of change in Hb will be measured by CBC at 6 weeks, 3 months, 6 months, and 1 year of enrollment.

SECONDARY OUTCOMES:
change in renal function (eGFR) | 6 weeks to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anita Mehrotra, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280